CLINICAL TRIAL: NCT00785252
Title: Randomized Study of the EZIO Compared to Central Venous Lines Used for Emergency Vascular Access
Brief Title: EZIO Compared to Central Venous Lines for Emergency Vascular Access
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor termination
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100731 (completed)
Record Dates: First submitted 2008-11-03; First posted 2008-11-05 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Catheters, Indwelling; Central Venous Line; Intraosseous Needle
Keywords: Catheters, Indwelling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): EZIO
  Interventions: Device: Powered Intraosseous device (EZIO)
- 2 (Experimental): Central line
  Interventions: Device: standard central line

INTERVENTIONS:
Device: Powered Intraosseous device (EZIO) — EZIO
  Arms: 1
Device: standard central line — placement of a central line
  Arms: 2

SUMMARY:
Multicenter randomized study to compare powered intraosseous access to standard central line access for the administration of fluids and drugs for patients in the Emergency Dept.

ELIGIBILITY:
Inclusion Criteria:

Over 18 years old Requires central access after peripheral access attempts have failed or are not otherwise feasible

Exclusion Criteria:

Fracture in target bone Not able to sign informed consent Excessive tissue or absence of adequate anatomical landmarks Known or suspected coagulopathies Pregnancy Patients in custody Patients with suspected great vessel injury Not fluid in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Time taken to place the device | ED visit

SECONDARY OUTCOMES:
Incidence of complications | ED visit
Costs for each of the two methods | Ed visit

CONTACTS AND LOCATIONS:
Overall Officials: Jeremty Brown, MD, Principal Investigator — George Washington University; Jeremy Brown, Principal Investigator — Dept of Emergency Medicine, GWU
Locations (1):
- Dept of Emergency Medicine, The George Washington University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- See also: Related Info — http://www.vidacare.com/